CLINICAL TRIAL: NCT00853099
Title: A Multi-Center, Randomized, Double-Blind, Placebo-controlled Study of Adalimumab in Japanese Subjects With Moderately to Severely Active Ulcerative Colitis.
Brief Title: A Study of Adalimumab in Japanese Subjects With Moderately to Severely Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10-447
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2012-11-27 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injections every 2 weeks for 52 weeks. From Week 8, participants with an inadequate response could switch to rescue therapy, where they initially received adalimumab 160 mg, 80 mg 2 weeks later, and then 40 mg every other week. Participants who completed the 52-week double-blind period received open-label adalimumab 40 mg every other week, with the possibility to escalate to 80 mg every other week, until drug approval.
  Interventions: Biological: adalimumab; Drug: placebo
- Adalimumab 80 mg/40 mg (Experimental): Participants received adalimumab 80 mg on Day 1, 40 mg at Week 2 and 40 mg every other week from Week 4 to Week 50, via subcutaneous injection. From Week 8, participants with an inadequate response could switch to rescue therapy, where they received adalimumab 40 mg every other week. Participants who completed the 52-week double-blind period received open-label adalimumab 40 mg every other week, with the possibility to escalate to 80 mg every other week, until drug approval.
  Interventions: Biological: adalimumab
- Adalimumab 160 mg/80 mg (Experimental): Participants received adalimumab 160 mg on Day 1, 80 mg at Week 2 and 40 mg every other week from Week 4 to Week 50, via subcutaneous injection. From Week 8, participants with an inadequate response could switch to rescue therapy, where they received adalimumab 40 mg every other week. Participants who completed the 52-week double-blind period received open-label adalimumab 40 mg every other week, with the possibility to escalate to 80 mg every other week, until drug approval.
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab
  Other Names: ABT-D2E7 Humira
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of adalimumab in Japanese subjects with moderately to severely active ulcerative colitis (UC).

DETAILED DESCRIPTION:
Patients who meet all of the inclusion criteria and none of the exclusion criteria are randomized 1:1:1 to receive subcutaneous injections of adalimumab at either 160/80 mg at Week 0/2 and 40 mg every other week (eow) starting at Week 4 to Week 50, 80/40 mg at Week 0/2 and 40 mg eow starting at Week 4 to Week 50, or placebo eow starting at Week 0 to Week 50 under the double-blind condition. At or after Week 8, participants who have inadequate response during the double-blind period can switch to the rescue arm, where participants from the placebo group initially receive adalimumab 160 mg and 80 mg 2 weeks later and those from the adalimumab group receive adalimumab 40 mg initially and 2 weeks later under double-blind conditions. All participants in the rescue arm then receive 40 mg adalimumab eow until Week 50. Participants who complete the 52-week double-blind period receive open-label adalimumab 40 mg eow starting at Week 52 and continuing until the end of the study. Participants who have an inadequate response or disease flare can dose escalate to 80 mg eow at or after Week 60. Participants who dose escalate to 80 mg eow and continue to have an inadequate response or disease flare are withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis for greater than 90 days prior to Baseline.
* Active ulcerative colitis with a Mayo Score of 6-12 points at Baseline and endoscopy subscore of 2-3 during the Screening Period, despite concurrent treatment with at least one of the following (oral corticosteroids or immunosuppressants or both as defined below):
* Stable oral corticosteroid dose (prednisolone dose of ≥ 20 mg/day or equivalent) for at least 14 days prior to Baseline or stable oral corticosteroid dose (prednisolone of 5 to less than 20 mg/day) for at least 40 days prior to Baseline. And/or
* At least a consecutive 90-day course of azathioprine or 6-mercaptopurine (6-MP) prior to Baseline, with a dose of azathioprine ≥ 50 mg/day or 6-MP ≥ 30 mg/day, or a dose that was the highest tolerated by the patient.

Exclusion Criteria:

* History of subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Koch pouch, or ileostomy for ulcerative colitis or was planning bowel surgery.
* Patients with disease limited to the rectum.
* Indeterminate colitis and/or Crohn's disease.
* Received any biological therapy (including infliximab) in the past.
* History of tuberculosis or malignancy.
* Pregnant women.
* Patients with positive C. difficile stool assay at Screening.
* Current diagnosis of fulminant colitis and/or toxic megacolon.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morio Ozawa, MS, Study Director — AbbVie
Locations (65):
- Japan (65):
  - Site Reference ID/Investigator# 47136, Asahikawa
  - Site Reference ID/Investigator# 47159, Chiba
  - Site Reference ID/Investigator# 47183, Chikushino-shi
  - Site Reference ID/Investigator# 47135, Fukuoka
  - Site Reference ID/Investigator# 47182, Fukuoka
  - Site Reference ID/Investigator# 47124, Hamamatsu
  - Site Reference ID/Investigator# 47130, Hirakata-shi
  - Site Reference ID/Investigator# 47103, Hirosaki
  - Site Reference ID/Investigator# 47131, Hiroshima
  - Site Reference ID/Investigator# 47178, Hiroshima
  - Site Reference ID/Investigator# 47179, Hiroshima
  - Site Reference ID/Investigator# 47176, Izumo
  - Site Reference ID/Investigator# 47226, Kagoshima
  - Site Reference ID/Investigator# 47123, Kanazawa
  - Site Reference ID/Investigator# 47160, Kashiwa
  - Site Reference ID/Investigator# 47108, Kawagoe
  - Site Reference ID/Investigator# 47107, Koshigaya
  - Site Reference ID/Investigator# 47181, Kurume
  - Site Reference ID/Investigator# 47222, Kurume
  - Site Reference ID/Investigator# 47223, Kurume
  - Site Reference ID/Investigator# 47127, Kyoto
  - Site Reference ID/Investigator# 47170, Kyoto
  - Site Reference ID/Investigator# 47171, Kyoto
  - Site Reference ID/Investigator# 47172, Kyoto
  - Site Reference ID/Investigator# 47134, Matsuyama
  - Site Reference ID/Investigator# 47225, Miyazaki
  - Site Reference ID/Investigator# 47138, Morioka
  - Site Reference ID/Investigator# 47168, Nagakute-shi
  - Site Reference ID/Investigator# 47125, Nagoya
  - Site Reference ID/Investigator# 47126, Nagoya
  - Site Reference ID/Investigator# 47166, Nagoya
  - Site Reference ID/Investigator# 47122, Niigata
  - Site Reference ID/Investigator# 47227, Nishihara
  - Site Reference ID/Investigator# 47174, Nishinomiya-shi
  - Site Reference ID/Investigator# 47177, Okayama
  - Site Reference ID/Investigator# 47228, Okinawa
  - Site Reference ID/Investigator# 47128, Osaka
  - Site Reference ID/Investigator# 47129, Osaka
  - Site Reference ID/Investigator# 47224, Ōita
  - Site Reference ID/Investigator# 47169, Ōtsu
  - Site Reference ID/Investigator# 47118, Sagamihara-shi
  - Site Reference ID/Investigator# 47158, Saitama-shi
  - Site Reference ID/Investigator# 47109, Sakura
  - Site Reference ID/Investigator# 15853, Sapporo
  - Site Reference ID/Investigator# 47137, Sapporo
  - Site Reference ID/Investigator# 47104, Sendai
  - Site Reference ID/Investigator# 47147, Sendai
  - Site Reference ID/Investigator# 47180, Susaki-shi
  - Site Reference ID/Investigator# 47133, Takamatsu
  - Site Reference ID/Investigator# 47173, Takatsuki-shi
  - Site Reference ID/Investigator# 47106, Tokorozawa-shi
  - Site Reference ID/Investigator# 47132, Tokushima
  - Site Reference ID/Investigator# 47110, Tokyo
  - Site Reference ID/Investigator# 47111, Tokyo
  - Site Reference ID/Investigator# 47112, Tokyo
  - Site Reference ID/Investigator# 47116, Tokyo
  - Site Reference ID/Investigator# 47117, Tokyo
  - Site Reference ID/Investigator# 47161, Tokyo
  - Site Reference ID/Investigator# 47164, Tokyo
  - Site Reference ID/Investigator# 47165, Toyama
  - Site Reference ID/Investigator# 47167, Toyoake
  - Site Reference ID/Investigator# 47105, Yamagata
  - Site Reference ID/Investigator# 47175, Yamatotakada
  - Site Reference ID/Investigator# 47120, Yokohama
  - Site Reference ID/Investigator# 47121, Yokohama

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Double-blind Placebo: Participants received placebo subcutaneous injections every 2 weeks for 52 weeks. From Week 8, participants with an inadequate response could switch to rescue therapy, where they initially received adalimumab 160 mg, 80 mg 2 weeks later, and then 40 mg every other week.
- Double-blind Adalimumab 80 mg/40 mg: Participants received adalimumab 80 mg on Day 1, 40 mg at Week 2 and 40 mg every other week from Week 4 to Week 50, via subcutaneous injection. From Week 8, participants with an inadequate response could switch to rescue therapy, where they received adalimumab 40 mg every other week.
- Double-blind Adalimumab 160 mg/80 mg: Participants received adalimumab 160 mg on Day 1, 80 mg at Week 2 and 40 mg every other week from Week 4 to Week 50, via subcutaneous injection. From Week 8, participants with an inadequate response could switch to rescue therapy, where they received adalimumab 40 mg every other week.
- All Adalimumab: All participants who received at least one dose of adalimumab during the study (adalimumab treatment groups in the double-blind phase, and participants randomized to placebo who received adalimumab in the rescue phase or open-label phase).
Period: Double-blind Period
Arm/Group | Double-blind Placebo | Double-blind Adalimumab 80 mg/40 mg | Double-blind Adalimumab 160 mg/80 mg | All Adalimumab
Started | 96 | 87 | 91 | 0
Treated | 96 | 87 | 90 (1 participant, incorrectly treated with open-label (rescue) study drug at Week 0, was excluded.) | 0
Completed Week 8 | 92 | 85 | 86 | 0
Completed | 73 (Participants who completed Week 52.) | 58 (Participants who completed Week 52.) | 60 (Participants who completed Week 52.) | 0
Not Completed | 23 | 29 | 31 | 0
Not completed — Adverse Event | 7 | 9 | 13 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 0
Not completed — Lack of Efficacy | 14 | 17 | 16 | 0
Not completed — Other | 0 | 0 | 1 | 0
Not completed — Mistreated with rescue study drug | 0 | 0 | 1 | 0
Period: Double-blind + Open-label Periods
Arm/Group | Double-blind Placebo | Double-blind Adalimumab 80 mg/40 mg | Double-blind Adalimumab 160 mg/80 mg | All Adalimumab
Started | 0 | 0 | 0 | 266 (7 participants randomized to placebo did not receive any adalimumab; 1 participant was excluded.)
Completed | 0 | 0 | 0 | 119
Not Completed | 0 | 0 | 0 | 147
Not completed — Lack of Efficacy | 0 | 0 | 0 | 74
Not completed — Adverse Event | 0 | 0 | 0 | 47
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 20
Not completed — Other | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: 1 participant in the adalimumab 160 mg/80 mg arm was incorrectly treated with open-label (rescue) study drug at Week 0, and was not included in Baseline Characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab 80 mg/40 mg | Adalimumab 160 mg/80 mg | Total
Number analyzed (Participants) | 96 | 87 | 90 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] — Demographic data are provided for the Full Analysis Set (participants who received at least one dose of study drug in the double-blind portion of the study).
  years | 41.3 (13.56) | 44.4 (15.04) | 42.5 (14.56) | 42.7 (14.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 37 | 29 | 92
  Male | 70 | 50 | 61 | 181
Region of Enrollment [Number; unit: participants]
  Japan | 96 | 87 | 90 | 273
Mayo score [Mean (Standard Deviation); unit: scores on a scale] — A composite score of ulcerative colitis disease activity calculated as the sum of 4 subscores:
  * Stool frequency, based on the participant's diary, scored from 0 (normal number of stools) to 3 (≥5 stools than normal);
  * Rectal bleeding, based on the participant's diary, scored from 0 (no blood) to 3 (blood only passed);
  * Endoscopy, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration);
  * Physician's Global Assessment, scored from 0 (normal) to 3 (severe disease). The total Mayo score ranges from 0 to 12; higher scores indicate more severe disease.
  scores on a scale | 8.5 (1.56) | 8.5 (1.42) | 8.6 (1.44) | 8.5 (1.47)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Remission at 8 Weeks
Description: Clinical remission was defined as a Mayo score ≤ 2 with no individual subscore > 1. The Mayo score is a composite score of ulcerative colitis disease activity calculated as the sum of four subscores:
  * Stool Frequency Subscore (SFS), based on the participant's diary and scored from zero (normal number of stools) to three (5 or more stools than normal);
  * Rectal Bleeding Subscore (RBS), based on the participant's diary and scored from zero (no blood) to three (blood only passed);
  * Endoscopy Subscore (ESS), based on colonoscopy or sigmoidoscopy and scored from zero (normal or inactive disease) to three (severe disease, spontaneous bleeding, ulceration);
  * Physician's Global Assessment (PGA) subscore, based on the physician's overall assessment, and scored from zero (normal) to three (severe disease).
  The total Mayo score ranges from 0 to 12 points, with higher scores representing more severe disease.
Time Frame: Week 8
Population: The full analysis set includes all patients who received at least 1 dose of study drug any time during the first 52 weeks and with at least 1 efficacy measurement after the first dose of study medication. Non-responder imputation (NRI) was used, where all missing values and values after the start of rescue treatment were considered non-remission.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab 80 mg/40 mg | Adalimumab 160 mg/80 mg
Number analyzed (Participants) | 96 | 87 | 90
percentage of participants | 11.5 | 13.8 | 10.0

2. Primary Outcome: Percentage of Participants With Clinical Remission at 52 Weeks
Description: as for outcome 1
Time Frame: Week 52
Population: Full analysis set. Non-responder imputation (NRI) was used, where all missing remission values and values after the start of rescue treatment were considered as non-remission.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab 80 mg/40 mg | Adalimumab 160 mg/80 mg
Number analyzed (Participants) | 96 | 87 | 90
percentage of participants | 7.3 | 26.4 | 20.0

3. Secondary Outcome: Percentage of Participants With Clinical Remission at 8, 32, and 52 Weeks
Description: Clinical remission was defined as a Mayo score ≤ 2 with no individual subscore > 1. The Mayo score is a composite score of ulcerative colitis disease activity calculated as the sum of four subscores:
  * Stool Frequency Subscore (SFS), based on the participant's diary and scored from zero (normal number of stools) to three (5 or more stools than normal);
  * Rectal Bleeding Subscore (RBS), based on the participant's diary and scored from zero (no blood) to three (blood only passed);
  * Endoscopy Subscore (ESS), based on colonoscopy or sigmoidoscopy and scores from zero (normal or inactive disease) to three (severe disease, spontaneous bleeding, ulceration);
  * Physician's Global Assessment (PGA) subscore, based on the physician's overall assessment, and scored from zero (normal) to three (severe disease).
  The total Mayo score ranges from 0 to 12 points, with higher scores representing more severe disease.
Time Frame: Weeks 8, 32, and 52
Population: Full analysis set, non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab 80 mg/40 mg | Adalimumab 160 mg/80 mg
Number analyzed (Participants) | 96 | 87 | 90
percentage of participants
  Week 8 | 11.5 | 13.8 | 10.0
  Week 32 | 8.3 | 17.2 | 17.8
  Week 52 | 7.3 | 26.4 | 20.0

4. Secondary Outcome: Percentage of Participants With a Clinical Response
Description: A clinical response was defined as a decrease in Mayo score of ≥ 3 points and ≥ 30% from Baseline PLUS a decrease in the Rectal Bleeding Subscore (RBS) ≥ 1 or an absolute RBS of 0 or 1.
  The Mayo score is a composite score of ulcerative colitis disease activity calculated as the sum of four subscores:
  * Stool Frequency Subscore, based on the participant's diary and scored from zero (normal number of stools) to three (5 or more stools than normal);
  * Rectal Bleeding Subscore, based on the participant's diary and scored from zero (no blood) to three (blood only passed);
  * Endoscopy Subscore, based on colonoscopy or sigmoidoscopy and scored from zero (normal or inactive disease) to three (severe disease, spontaneous bleeding, ulceration);
  * Physician's Global Assessment subscore, based on the physician's overall assessment, and scored from zero (normal) to three (severe disease).
  The total Mayo score ranges from 0 to 12 points, with higher scores representing more severe disease.
Time Frame: Baseline and Weeks 8, 32, and 52
Population: Full analysis set, non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab 80 mg/40 mg | Adalimumab 160 mg/80 mg
Number analyzed (Participants) | 96 | 87 | 90
percentage of participants
  Week 8 | 35.4 | 42.5 | 50.0
  Week 32 | 20.8 | 33.3 | 37.8
  Week 52 | 17.7 | 29.9 | 31.1

5. Secondary Outcome: Percentage of Participants With Mucosal Healing
Description: Mucosal healing was defined as an endoscopy subscore of ≤ 1 and was assessed using flexible sigmoidoscopy performed at Weeks 8, 32, and 52.
  The endoscopy subscore ranges from zero to three as follows:
  0 = Normal or inactive disease, 1 = Mild disease (erythema, decreased vascular pattern, mild friability), 2 = Moderate disease (marked erythema, absent vascular pattern, friability, erosions), 3 = Severe disease (spontaneous bleeding, ulceration).
Time Frame: Weeks 8, 32, and 52
Population: Full analysis set, non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab 80 mg/40 mg | Adalimumab 160 mg/80 mg
Number analyzed (Participants) | 96 | 87 | 90
percentage of participants
  Week 8 | 30.2 | 39.1 | 44.4
  Week 32 | 21.9 | 27.6 | 31.1
  Week 52 | 15.6 | 28.7 | 28.9

6. Secondary Outcome: Percentage of Participants With Rectal Bleeding Subscore Indicative of Mild Disease (≤ 1)
Description: Rectal bleeding was assessed from the participant's diary, taking the worst score from the 3 days prior to each study visit. The rectal bleeding subscore ranges from zero to three, according to the following scale:
  0 = no blood seen, 1 = streaks of blood with stool less than half the time, 2 = obvious blood with stool most of the time, 3 = blood alone passed.
Time Frame: Weeks 8, 32, and 52
Population: Full analysis set, non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab 80 mg/40 mg | Adalimumab 160 mg/80 mg
Number analyzed (Participants) | 96 | 87 | 90
percentage of participants
  Week 8 | 67.7 | 80.5 | 71.1
  Week 32 | 28.1 | 40.2 | 43.3
  Week 52 | 22.9 | 32.2 | 34.4

7. Secondary Outcome: Percentage of Participants With Physician's Global Assessment Subscore Indicative of Mild Disease (≤ 1)
Description: The Physician's Global Assessment Subscore acknowledges the three other subscores (Stool Frequency, Rectal Bleeding, and Endoscopy), the participant's daily record of abdominal discomfort and functional assessment, and other observations such as physical findings and the participant's performance status. Possible scores range from zero to three as follows:
  0 = Normal (other subscores are 0), 1 = Mild disease (other subscores are mostly 1), 2 = Moderate disease (other subscores are 1 to 2), 3 = Severe disease (other subscores are 2 to 3).
Time Frame: Weeks 8, 32, and 52
Population: Full analysis set, non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab 80 mg/40 mg | Adalimumab 160 mg/80 mg
Number analyzed (Participants) | 96 | 87 | 90
percentage of participants
  Week 8 | 44.8 | 47.1 | 61.1
  Week 32 | 28.1 | 36.8 | 37.8
  Week 52 | 19.8 | 29.9 | 34.4

8. Secondary Outcome: Percentage of Participants With Stool Frequency Subscore Indicative of Mild Disease (≤ 1)
Description: Stool frequency was assessed from the participant's diary, taking the worst score from the 3 days prior to each study visit. The stool frequency subscore ranges from zero to three, according to the following scale:
  0 = Normal number of stools for this participant, 1 = 1-2 stools more than normal, 2 = 3-4 stools more than normal, 3 = 5 or more stools more than normal.
Time Frame: Weeks 8, 32, and 52
Population: Full analysis set, non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab 80 mg/40 mg | Adalimumab 160 mg/80 mg
Number analyzed (Participants) | 96 | 87 | 90
percentage of participants
  Week 8 | 32.3 | 34.5 | 40.0
  Week 32 | 20.8 | 33.3 | 31.1
  Week 52 | 13.5 | 28.7 | 28.9

9. Secondary Outcome: Percentage of Inflammatory Bowel Disease Questionnaire (IBDQ) Responders
Description: An inflammatory bowel disease questionnaire responder was defined as a participant with at least a 16-point increase from Baseline in total Inflammatory Bowel Disease Questionnaire (IBDQ) score. The IBDQ is a 32-item questionnaire consisting of 4 dimensions: bowel-related symptoms, systemic function, social function, and emotional status. The responses to each question within each domain range from 1 (significant impairment) to 7 (no impairment), with the total score ranging from 32 (very poor) to 224 (perfect health-related quality of life).
Time Frame: Baseline and Weeks 8, 32, and 52
Population: Full analysis set, non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab 80 mg/40 mg | Adalimumab 160 mg/80 mg
Number analyzed (Participants) | 96 | 87 | 90
percentage of participants
  Week 8 | 39.6 | 48.3 | 42.2
  Week 32 | 21.9 | 33.3 | 28.9
  Week 52 | 12.5 | 29.9 | 21.1

10. Secondary Outcome: Number of Participants With Adverse Events up to Week 8
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
  The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related.
  A serious adverse event is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
  For more details on adverse events please see the Adverse Event section below.
Time Frame: 8 weeks
Population: The Safety Analysis Set includes all participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Adalimumab 80 mg/40 mg | Adalimumab 160 mg/80 mg
Number analyzed (Participants) | 96 | 87 | 90
participants
  Any adverse event | 45 | 49 | 40
  Any AE at least possibly drug related | 10 | 14 | 12
  Any serious adverse event | 7 | 2 | 4
  Any AE leading to discontinuation of study drug | 4 | 0 | 6

11. Secondary Outcome: Number of Participants With Adverse Events up to Week 52
Description: as for outcome 10
Time Frame: 52 weeks
Population: The safety analysis set.
Measure: Number; unit: participants
Arm/Group | Placebo | Adalimumab 80 mg/40 mg | Adalimumab 160 mg/80 mg
Number analyzed (Participants) | 96 | 87 | 90
participants
  Any adverse event | 67 | 68 | 75
  Any AE at least possibly drug related | 17 | 23 | 32
  Any serious adverse event | 12 | 14 | 10
  Any AE leading to discontinuation of study drug | 5 | 5 | 12

12. Secondary Outcome: Number of Participants With Adverse Events During the Adalimumab Treatment Period
Description: as for outcome 10
Time Frame: 221 weeks
Population: The safety analysis set.
Measure: Number; unit: participants
Arm/Group | All Adalimumab
Number analyzed (Participants) | 266
participants
  Any adverse event | 261
  Any AE at least possibly drug related | 142
  Any serious adverse event | 90
  Any AE leading to discontinuation of study drug | 37

ADVERSE EVENTS:
Time Frame: For the 3 randomized treatment arms, adverse events (AEs) were reported from the time of study drug administration up to Week 52 (double-blind period); for All Adalimumab, AEs were reported up to 221 weeks+70 days following discontinuation of study drug.
Description: Serious AEs (SAEs) were collected from the time participants signed the study-specific informed consent. For SAEs, the number of participants affected in the Double-blind Placebo arm (n=13) is reported from the final database lock, versus the number reported in Outcome Measure 11 (n=12), which was from the interim database lock.
Arm/Group | Double-blind Placebo | Double-blind Adalimumab 80 mg/40 mg | Double-blind Adalimumab 160 mg/80 mg | All Adalimumab
Serious Adverse Events (participants affected / at risk) | 13/96 | 14/87 | 10/90 | 90/266
Other Adverse Events (participants affected / at risk) | 51/96 | 47/87 | 60/90 | 235/266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=96) | Double-blind Adalimumab 80 mg/40 mg (N=87) | Double-blind Adalimumab 160 mg/80 mg (N=90) | All Adalimumab (N=266)
ATRIAL FLUTTER (Cardiac disorders) | 0 | 0 | 1 | 1
PERICARDITIS (Cardiac disorders) | 0 | 0 | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
DIABETIC RETINOPATHY (Eye disorders) | 0 | 0 | 0 | 1
COLITIS ULCERATIVE (Gastrointestinal disorders) | 8 | 5 | 5 | 38
COLONIC POLYP (Gastrointestinal disorders) | 0 | 1 | 0 | 3
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GASTROINTESTINAL DYSPLASIA (Gastrointestinal disorders) | 0 | 0 | 1 | 3
INTESTINAL POLYP (Gastrointestinal disorders) | 0 | 0 | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
RECTAL STENOSIS (Gastrointestinal disorders) | 1 | 0 | 0 | 1
RECTAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ADVERSE DRUG REACTION (General disorders) | 0 | 1 | 0 | 1
DEATH (General disorders) | 0 | 0 | 1 | 1
DRUG INTOLERANCE (General disorders) | 0 | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 0 | 1
MALAISE (General disorders) | 0 | 0 | 0 | 2
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 2
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1
APPENDICITIS (Infections and infestations) | 0 | 0 | 0 | 1
BACTERIAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 1 | 2
BURSITIS INFECTIVE (Infections and infestations) | 0 | 0 | 0 | 1
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
ENTERITIS INFECTIOUS (Infections and infestations) | 1 | 0 | 0 | 2
ERYSIPELAS (Infections and infestations) | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 2
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
GINGIVITIS (Infections and infestations) | 0 | 0 | 1 | 1
INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
PELVIC ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 1
PNEUMONIA BACTERIAL (Infections and infestations) | 0 | 1 | 1 | 3
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 0 | 0 | 0 | 1
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 1 | 0 | 2
TUBERCULOSIS (Infections and infestations) | 0 | 0 | 1 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
HEAT ILLNESS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
WOUND (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
DRUG LEVEL (Investigations) | 0 | 1 | 0 | 1
MEDICAL OBSERVATION (Investigations) | 0 | 0 | 0 | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
PARATHYROID TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 0 | 1
EPILEPSY (Nervous system disorders) | 0 | 0 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 1 | 0 | 1
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 0 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 1
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 0 | 0 | 0 | 1
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
IMMUNOSUPPRESSANT DRUG THERAPY (Surgical and medical procedures) | 0 | 0 | 0 | 1
TAKAYASU'S ARTERITIS (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=96) | Double-blind Adalimumab 80 mg/40 mg (N=87) | Double-blind Adalimumab 160 mg/80 mg (N=90) | All Adalimumab (N=266)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 7 | 4 | 8 | 24
COLITIS ULCERATIVE (Gastrointestinal disorders) | 5 | 2 | 5 | 20
DENTAL CARIES (Gastrointestinal disorders) | 5 | 6 | 3 | 27
NAUSEA (Gastrointestinal disorders) | 4 | 2 | 5 | 26
STOMATITIS (Gastrointestinal disorders) | 1 | 0 | 1 | 14
VOMITING (Gastrointestinal disorders) | 1 | 0 | 4 | 23
INJECTION SITE REACTION (General disorders) | 2 | 7 | 6 | 25
MALAISE (General disorders) | 0 | 3 | 7 | 13
PYREXIA (General disorders) | 4 | 4 | 5 | 24
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 | 1 | 1 | 14
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 2 | 16
INFLUENZA (Infections and infestations) | 6 | 3 | 4 | 20
NASOPHARYNGITIS (Infections and infestations) | 21 | 19 | 30 | 162
ORAL HERPES (Infections and infestations) | 0 | 1 | 0 | 14
PHARYNGITIS (Infections and infestations) | 2 | 1 | 1 | 15
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2 | 3 | 6 | 22
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 21
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4 | 31
HEADACHE (Nervous system disorders) | 6 | 3 | 7 | 42
INSOMNIA (Psychiatric disorders) | 2 | 2 | 3 | 23
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 23
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 5 | 27
ECZEMA (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 27
RASH (Skin and subcutaneous tissue disorders) | 5 | 4 | 3 | 27
HYPERTENSION (Vascular disorders) | 2 | 1 | 1 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.